CLINICAL TRIAL: NCT01487239
Title: A Phase I Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-GDC-0980 Following Single Oral Dose Administration in Healthy Postmenopausal Female Subjects
Brief Title: Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-GDC-0980 Following Single Oral Dose Administration in Healthy Postmenopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP27915
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (1):
- A (Experimental): [14C]-GDC-0980 administered as a 10-mg oral dose
  Interventions: Drug: [14C]-GDC-0980

INTERVENTIONS:
Drug: [14C]-GDC-0980 — 100 uCi of [14C]-GDC-0980 in total dose of 10 mg GDC-0980

SUMMARY:
This study will be an open-label, non-randomized, absorption, metabolism, and excretion study of [14C]-GDC-0980 administered as a 10-mg oral dose to 6 healthy postmenopausal and/or surgically sterile female subjects following at least a 10-hour fast from food (not including water).

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy as determined by the absence of clinically significant findings in the medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator
* Female subjects of non-childbearing potential, as defined as either: postmenopausal and without recent history of menorrhea as documented either by physician note or confirmed by serum follicle-stimulating hormone level consistent with postmenopausal status, or surgically sterile
* BMI range within 18.5 to 29.9 kg/m2, inclusive
* Negative test for selected drugs of abuse at Screening and at Check-in
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg], hepatitis C virus antibody [anti-HCV] and negative HIV antibody screens
* Minimum of 1 to 2 bowel movements per day

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* History or presence of inflammatory diseases, including those with small or large intestine inflammation such as Crohn's disease or ulcerative colitis, which required immunosuppressants
* Use of potent proton-pump inhibitors such as omeprazole, lansoprazole, dexlansoprazole, esomeprazole, pantoprazole, and rabeprazole
* History of Gilbert's Syndrome
* History of diabetes mellitus and/or elevated fasting glucose at baseline
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction within 1 year prior to Check-in
* Participation in more than one other radiolabeled investigational study drug trial within 12 months prior to Check-in. The previous radiolabeled study drug must have been received more than 6 months prior to Check-in for this study and the total exposure from this study and the previous study will be within the recommended levels considered safe
* Exposure to significant radiation 12 months prior to Check-in
* Use of any tobacco-containing or nicotine-containing products within 3 months/approximately 90 days prior to Check-in or positive urine screening for cotinine
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Check-in
* Use of any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator
* Use of any over-the-counter (OTC), non-prescription preparations within 7 days prior to Check-in
* Use of alcohol-, grapefruit-, or caffeine-containing foods or beverages within 72 hours
* Poor peripheral venous access
* Donation of blood from 30 days prior to Screening or of plasma from 2 weeks prior to Screening
* Receipt of blood products within 2 months prior to Check-in
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: maximum observed concentration (Cmax) | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: time to maximum concentration (tmax) | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: area under the concentration-time curve from Hour 0 to the last measurable concentration (AUC0-t) | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: area under the concentration-time curve extrapolated to infinity | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: apparent terminal elimination half-life (t1/2) | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: apparent terminal phase elimination rate constant | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: apparent total clearance | up to approximately 5 weeks
Pharmacokinetic based on the plasma concentrations of total radioactivity and GDC-0980: apparent volume of distribution | up to approximately 5 weeks

SECONDARY OUTCOMES:
Pharmacokinetic based on the urine radioactivity concentrations: amount of drug excreted in the urine over sampling interval | up to approximately 5 weeks
Pharmacokinetic based on the urine radioactivity concentrations: renal clearance | up to approximately 5 weeks
Pharmacokinetic based on the urine radioactivity concentrations: percent excreted in urine | up to approximately 5 weeks
Pharmacokinetic parameters for the metabolites of [14C]-GDC-0980 calculated based on plasma, urine, and fecal concentration levels. | up to approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Madison, Wisconsin, United States